CLINICAL TRIAL: NCT03478605
Title: Phase II Randomized Trial to Evaluate Efficacy of Olanzapine With Short-acting 5HT3 Inhibitors in Chemotherapy-induced Nausea & Vomiting (CINV) Prophylaxis
Brief Title: Trial to Evaluate Efficacy of Olanzapine With Short-acting 5HT3 Inhibitors in Chemotherapy-induced Nausea & Vomiting (CINV) Prophylaxis
Acronym: OlaCINV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Collaborators: RUSSCO/RakFond (Unknown)
Responsible Party: Principal Investigator, Alexey Rumyantsev, MD, Blokhin's Russian Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OlaCINV; 2018-01-YS-ECI (Other Grant/Funding Number: RUSSCO/RakFond)
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Emesis; Vomiting; Nausea Post Chemotherapy; Nausea; Chemotherapy-induced Nausea and Vomiting
Keywords: olanzapine; aprepitant; CINV; nausea; vomiting; nausea and vomiting; antiemetics
MeSH Terms: conditions — Vomiting; Nausea | interventions — Olanzapine; Aprepitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase II randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olanzapine (Experimental): Olanzapine 5 mg/day p.o. d 0-4 + ondansetron 16 mg IV d 1 + dexamethasone 12 mg IV d 1, 8 mg b.i.d.; IM or P.O. d 2-4;
  Interventions: Drug: Olanzapine; Drug: Ondansetron; Drug: Dexamethasone
- Aprepitant (Active Comparator): Aprepitant 125 mg p.o d 1 + 80 mg p.o d 2,3 + ondansetron 16 mg IV d 1 + dexamethasone 12 mg IV d 1, 8 mg b.i.d. IM or P.O. d 2-4;
  Interventions: Drug: Aprepitant Pill; Drug: Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 5 mg/day will be administered orally on days 0-4 of chemotherapy cycle (before bedtime)
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Aprepitant Pill — Aprepitant 125 mg orally will be administered on day 1 of chemotherapy cycle; 80 mg - on days 2 and 3.
  Other Names: Emend
  Arms: Aprepitant
Drug: Ondansetron — Ondansetron 16 mg IV on day 1 of chemotherapy cycle (as standard component of antiemetic therapy)
Drug: Dexamethasone — Dexamethasone 8 mg IV on day 1 of chemotherapy cycle; 8 mg IV or orally on days 2-3 (as standard component of antiemetic therapy)

SUMMARY:
Olanzapine-containing regimens for CINV prophylaxis may provide even better protection than aprepitant-containing regimens.

DETAILED DESCRIPTION:
Olanzapine-containing regimens for CINV provide high complete response (CR) rate in patients receiving high emetogenic chemotherapy. Olanzapine may be more effective than aprepitant in this setting but cheaper. However, there is no strong evidence supporting the advantages of olanzapine over aprepitant - and this is the reason why aprepitant is still the standard of care. Due to high cost aprepitant can be not affordable in low- and middle income countries; this compromises quality of life of cancer patients. On the other hand, recommended olanzapine-based regimen includes palonosetron, whose price is quite high as well and undesired sedation is a common side effect for olanzapine doses that currently recommended, these adverse events precludes wide use of olanzapine in oncology. Development of effective, tolerable and affordable regimen for CINV prophylaxis based on low-dose olanzapine and short-acting 5-HT3 inhibitors can improve quality of care for many cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. High-emetogenic chemotherapy (HEC) regimen (e.g., cisplatin ≥70 mg/m2 or doxorubicin ≥60 mg/m2 or carboplatin AUC≥4). Patients that are prescribed less doses of mentioned agents are still allowed if another high-emetogenic drug will be administered (eg, doxorubicin plus cisplatin);
2. Administration of HEC component only in first day of the cycle;
3. No previous chemotherapy or radiotherapy;
4. No concomitant quinolone antibiotics administration;
5. ECOG PS ≤2;
6. No nausea and vomiting 24 hours before enrollment;
7. Adequate hepatic and renal function (eg, ALaT, ASaT ≤3 ULN, creatinine clearance ≥50 ml/minute).
8. No brain metastases, leptomeningeal carcinomatosis, and chronic diseases such as uncontrolled diabetes mellitus and chronic alcohol consumption.
9. Subject willing to participate in the trial and provided informed consent form.

Exclusion Criteria:

1. Previous chemotherapy or radiotherapy;
2. Moderate- or low- emetogenic chemotherapy;
3. Multiday administration of HEC agents;
4. ECOG PS >2;
5. History of brain metastases, signs of symptoms of bowel obstruction;
6. Nausea and/or vomiting of any genesis 24 hours before enrollment;
7. Uncontrolled diabetes mellitus or other metabolic diseases; chronic alcohol consumption.
8. Diseases and conditions interfere with subject ability to swallow the drug and to take oral medication;
9. Concomitant therapy with olanzapine or other antipsychotic drugs; history of mental illness;
10. Concomitant therapy with quinolone antibiotics;
11. Contraindications for olanzapine or aprepitant administration;
12. Intraperitoneal or intrapleural administration of HEC drugs;
13. Inadequate hepatic and/or renal function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-05-25 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Nausea control | 0-120 hours after chemotherapy
  Complete control of nausea (ie, no nausea) in overall treatment period (0-120 hours after chemotherapy).

SECONDARY OUTCOMES:
Complete Response Rate in Overall Treatment Period | 0-120 hours after chemotherapy
  Complete response rate (ie, no vomiting, no use of rescue medication) in 0-120 hours after chemotherapy
Rate of undesired sedation | 0-120 hours after chemotherapy
  Rate of undesired sedation 0-120 hours after chemotherapy
Complete Response Rate in Acute Treatment Period | 0-24 hours after chemotherapy
  Complete response rate (ie, no vomiting, no use of rescue medication) in 0-24 hours after chemotherapy
Complete Response Rate in Delayed Treatment Period | 24-120 hours after chemotherapy
  Complete response rate (ie, no vomiting, no use of rescue medication) in 24-120 hours after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Blokhin Cancer Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided